CLINICAL TRIAL: NCT03741738
Title: The Investigation on the Expression of High Mobility Group Protein Box-1 (HMGB1) in Peripheral Blood of Vitiligo Patients and Healthy Controls According to Clinical Features, Treatment and Disease Activity
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2018-0686
Record Dates: First submitted 2018-10-31; First posted 2018-11-15 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum of patient will be evaluated
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-segmental vitiligo :: A. Patients aged 19 years or older who were clinically diagnosed with non-segmented leukopenia at Severance Hospital.
  B. Patients (36 patients) who experienced worsening symptoms within the last 3 months and 10 patients whose symptoms were stable within 3 months C. Patients with vitiligo lesion at least 3% of the skin
- Segmental VT or Focal VT: A. The investigators evaluated patients who were diagnosed as segmental vitiligo clinically on Severance hospital and who were 19 years old or older.
- Normal control: A. Subjects aged 19 or older who do not have not only vitiligo but also other skin and systemic diseases

SUMMARY:
Vitiligo is an acquired depigmented disorder that causes white spots on the skin due to the loss of melanocytes. It is a common disease which accounts for 0.5-1% of the whole population. It is a refractory skin disease with 25-50 thousand patients in Korea. And it is often caused in the exposed areas of the patient, causing a great deal of mental and social dysfunction in the patient's life, and may lead to suicide attempts.

DETAILED DESCRIPTION:
A nationwide study conducted by the Korean Academy of vitiligo showed that 61.8% of patients with vitiligo always have emotional impairment. In addition, the incidence of recurrence is high, and the recurrence rate is reported up to 40% within one year after the discontinuation of treatment. Therefore, development of a marker for monitoring the disease activity is very important and desperately needed.

HMGB1 is a protein located in the nucleus, such as histone, and binds to genes and transcription factors to stabilize and control the DNA transcription. However, when released from the cells, it acts as a danger signal and is thought to cause autoimmune diseases such as inflammatory diseases and lupus. The present study demonstrated through ex vivo tissue culture that HMGB1 can induce melanocyte apoptosis by inducing apoptosis and also observed that serum concentration of HMGB1 was higher in vitiligo patients than in normal controls . The aim of this study is to investigate the usefulness of HMGB1 as a biomarker for predicting the severity of disease and to confirm the association between HMGB1 levels and vitiligo activity.

ELIGIBILITY:
Inclusion Criteria:

1. Non-segmental vitiligo :

   A. Patients aged 19 years or older who were clinically diagnosed with non-segmented leukopenia at Severance Hospital.

   B. Patients (36 patients) who experienced worsening symptoms within the last 3 months and 10 patients whose symptoms were stable within 3 months C. Patients with vitiligo lesion at least 3% of the skin
2. Segmental VT or Focal VT A. The investigators evaluated patients who were diagnosed as segmental vitiligo clinically on Severance hospital and who were 19 years old or older.
3. Normal control A. Subjects aged 19 or older who do not have not only vitiligo but also other skin and systemic diseases
4. Subjects who voluntarily signed a written consent before he / she fully explained the purpose and contents of the examination prior to clinical research
5. Subjects who can follow up during the clinical study

Exclusion Criteria:

1. Patients diagnosed with nevus depigmentosus in vitiligo group
2. Patients under the age of 19
3. Patients taking steroids and immunosuppressants within the last 4 weeks
4. Patients using steroids and immunomodulatory ointment within the last 2 weeks
5. Patients who have been treated with short-wave UV therapy and excimer laser within the last month
6. Subjects with a disease known to have elevated blood levels of HMGB1 (lupus, systemic cirrhosis Symptoms, infectious diseases, etc.) on normal group
7. Subjects do not want it or did not fill out a consent form
8. Subjects who are pregnant or lactating
9. Patients whose clinical investigator is deemed unsuitable as a subject for the following patients or other pathologies 1) If the site of treatment has infectious or inflammatory skin disease 2) If the site of treatment has melasma or other pigmented dermatologic disease 3) If subjects have keloid disease, collagen, or elastic fiber disease 4) If subjects have chronic wasting disease (asthma, diabetes, etc.) 5) If subjects are taking anticoagulants and are at risk of bleeding 6) If subjects have an autoimmune disease 7) Subjects with psychiatric problems 8) Acute patients
10. Others in addition to the above items, if it is deemed difficult for clinical practice to be conducted at the discretion of the clinical trial manager (including illiteracy and other foreigners exclusion)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who visted Severance hospital due to vitiligo
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2020-06-09 (Actual); Study Completion 2020-06-09 (Actual)

PRIMARY OUTCOMES:
Serum HMGB1 | Baseline
  Comparative analysis of serum HMGB1 between active non-segmental vitiligo and normal controls

SECONDARY OUTCOMES:
Serum HMGB1 | 3 months
  Analysis of serum HMGB1 between segmental vitiligo and normal control

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology, Severance Hospital, Cutaneous Biology Research Institute, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No